CLINICAL TRIAL: NCT05101733
Title: Pilot Study Regarding Mold Allergy in Austria: Clinical Relevance of Alternaria Alternata and Related Species
Brief Title: Mold Allergy in Austria: Clinical Relevance of Alternaria Alternata and Related Species
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Markus Berger, Dr. med. univ., Medical University of Vienna
Other Study IDs: 1318/2021
Record Dates: First submitted 2021-09-30; First posted 2021-11-01 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Fungal Allergy; Allergy
Keywords: Allergy; Fungal allergy; Alternaria alternata
MeSH Terms: conditions — Hypersensitivity | interventions — Nasal Provocation Tests; Patch Tests; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alternaria allergy sufferers: 50 people suffering from an allergy to Alternaria. These participants receive a questionnaire, a Skin-Prick-Test, a blood draw and nasal provocation with collection of nasal secretion
  Interventions: Diagnostic Test: Nasal provocation; Diagnostic Test: Skin-Prick Test; Diagnostic Test: Blood draw; Diagnostic Test: Collection of nasal secretion
- Non-allergic participants: Non allergic participants (20) receive a questionnaire, a blood draw and collection of nasal secretion
  Interventions: Diagnostic Test: Blood draw; Diagnostic Test: Collection of nasal secretion

INTERVENTIONS:
Diagnostic Test: Nasal provocation — Nasal provocation with Alternaria alternata extract. Changes in nasal mucosa are measured with a rhinomanometry device
  Groups: Alternaria allergy sufferers
Diagnostic Test: Skin-Prick Test — Skin-Prick-Test is administered to determine an allergy against Alternaria
  Groups: Alternaria allergy sufferers
Diagnostic Test: Blood draw — For further analysis
Diagnostic Test: Collection of nasal secretion — Allergy sufferers: After nasal provocation Non-allergics: After administration of isotonic nasal spray

SUMMARY:
Mold allergies are becoming increasingly important among the population. Increasing amounts of fungal spores are analyzed in air-samples because of urbanization, industrialization of food products and climate change. Mold also grows indoor and hence lead to additional health complaints.

Alternaria alternata, and its only major allergen Alt a 1, is the most important fungus for allergy sufferers. Alternaria alternata can not only cause allergic symptoms but can also cause intensified asthmatic symptoms.

Besides Alternaria alternata, there are over 700 other species of the genus Alternaria. The influence of these other species on allergic symptoms is poorly understood.

Furthermore, prevalence and incidence of an allergy to Alternaria alternata among the Austrian population is not known. Estimates range between 1-5% among the Austrian population.

This study aims to further investigate the incidence and characteristics of an allergy to Alternaria in Austria. This will be investigated with the help of participants (50 Alternaria allergy sufferers and 20 non allergic participants), spore counts in Austria and crowd-sourced symptom data.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be healthy people over 18 years of age. Allergic participants should have an allergic reaction against Alternaria, visible in the Skin-Prick-Test. Furthermore symptom data in the pollen diary of the Austrian Pollen Information Service should be existing

Exclusion Criteria:

* Subjects participating in a pharmacological study, pregnant subjects and subjects with an existing infectious- and/or autoimmune disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants are recruited with the help of advertisements on the social media pages of the Austrian Pollen Information Service and on the pollen diary app
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence, Immunoglobulin-E (IgE)-antibodies to selected Alternaria species | 12 months
  Determine the prevalence of sensitization to multiple Alternaria species in the Austrian population

SECONDARY OUTCOMES:
Cytokine-profile (e.g. Interleukin-13, Interleukin-5, Interleukin-10, TNFalpha, IFNgamma) upon Alt a 1 incubation | 12 months
  Changes in the immun response when ligand-binding mononuclear cells from the blood to Alt a 1, characterized by the cytokine profile (Th1/Th2/regulatory) and the cell population (B- and T-cells, macrophages/monocytes)

CONTACTS AND LOCATIONS:
Overall Officials: Erika Jensen-Jarolim, Univ.-Prof. Dr., Study Director — Department of Pathophysiology and Allergy Research
Locations (1):
- Medical University of Vienna, Vienna, Austria